CLINICAL TRIAL: NCT06586424
Title: The Prognostic Value of Anion Gap in Predicting Major Adverse Cardiovascular Events Among Patients With ST-Segment Elevation Myocardial Infarction
Acronym: ANGIO-STEMI
Status: Recruiting | Type: Observational
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Sodiqur Rifqi, Principal Investigator; Former of Head of Department of Cardiovascular Medicine Faculty of Medicine Universitas Diponegoro, Universitas Diponegoro
Other Study IDs: Undip_Kardio 2
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: anion gap; major adverse cardiovascular events; st-segment elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Acid-Base Equilibrium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MACE group: Patient with STEMI who suffered major adverse cardiovascular events (MACE) after underwent primary percutaneous coronary intervention (PPCI)
  Interventions: Diagnostic Test: Anion gap

INTERVENTIONS:
Diagnostic Test: Anion gap — Patient was taken blood examination before PPCI

SUMMARY:
This study aims to evaluate the prognostic value of the anion gap in predicting major adverse cardiovascular events among patients with ST-segment elevation myocardial infarction. Researchers will collect information based on hospital registry as secondary data of in patient who had diagnosed as ST-segment elevation myocardial infarction and underwent primary percutaneous coronary intervention. The data consist of demographic data, clinical presentation, laboratory, and angiography result were collected from hospital registry by reviewing medical record. Then, the data was analyzed by using IBM SPSS Statistics v26.

ELIGIBILITY:
Inclusion Criteria:

* Adults with 18 - 70 years old with diagnosis of STEMI who underwent PPCI

Exclusion Criteria:

* History of heart failure due to any causes
* Cardiogenic shock before PPCI
* Any infection at the time of presentation
* Pregnant woman
* Other causes of high anion gap levels such as chronic kidney disease, metabolic acidosis, etc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ST-segment elevation myocardial infarction who underwent PPCI
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | During hospitalization, up to 1 weeks

SECONDARY OUTCOMES:
Incidence of mortality | During hospitalization, up to 1 weeks
Incidence of reinfarction | During hospitalization, up to 1 weeks
Incidence of stroke | During hospitalization, up to 1 weeks
Incidence of lethal arrhythmia | During hospitalization, up to 1 weeks
Incidence of acute lung oedema | During hospitalization, up to 1 weeks
Incidence of cardiogenic shock | During hospitalization, up to 1 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No